CLINICAL TRIAL: NCT07373262
Title: Avacopan Added to Standard-of-care Therapy in ANCA-associated Vasculitis With Severe Kidney Involvement: a Randomized, Placebo-controlled, Double-blinded Multicenter Superiority Study
Brief Title: Avacopan Added to Standard-of-care Therapy in ANCA-associated Vasculitis With Severe Kidney Involvement
Acronym: REVERSE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC31/24/0321; 2024-519620-24-01 (EU CTIS Number)
Record Dates: First submitted 2025-12-23; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: ANCA-Associated Vasculitis (AAV)
Keywords: ANCA-associated vasculitis; avacopan
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — avacopan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GCs-based SOC + avacopan (Experimental): Patients will be standard of care (SOC and GCs) and receive Avacopan
  Interventions: Drug: Avacopan
- GCs-based SOC + placebo (Placebo Comparator): Patients will be standard of care (SOC and GCs) and receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avacopan — At day 0, and weeks 4, 8, 12, 20 36 patients will have avacopan dispensation
  Arms: GCs-based SOC + avacopan
Drug: Placebo — At day 0, and weeks 4, 8, 12, 20 36 patients will have placebo dispensation
  Arms: GCs-based SOC + placebo

SUMMARY:
ANCA-associated vasculitis (AAV) is a rare auto-immune disease, with high mortality in the absence of treatment. There is still an unmet need to define new treatment strategies to reduce drug side effects, as well as to reverse rare cases of refractory AAV and improve the kidney response to improve the long-term outcomes.

Severe forms of AAV-related necrotizing and crescentic rapidly progressive glomerulonephritis (RPGN) (i.e. estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m²) are associated with higher mortality, higher incidence of infections, and long-term consequences including chronic kidney disease (CKD) with subsequent complications (end-stage kidney disease (ESKD) requiring dialysis, cardiovascular diseases) and a burden of financial costs.

In patients with AAV and RPGN, recent guidelines recommend using a standard-of-care (SOC) immunosuppressive regimen including an induction regimen (rituximab or cyclophosphamide), plus glucocorticoids (GCs) (starting at 60 mg/day and tapering over 6-12 months) (+ or - plasma exchanges).

Since GCs also participate to the long-term control of AAV, new molecular pathophysiology-driven therapeutic approaches rapidly blocking and/or reversing AAV lesions are needed to go beyond the progressive control of AAV using GCs alone. Thus, an add-on approach including GCs-based immunosuppressive regimen plus a new targeted therapy may lead to both AAV control (systemic disease) and improvement of the kidney outcome (organ involvement).

Avacopan a selective inhibitor of the C5a receptor, recently emerged as a new therapeutic option in AAV. In a phase 3 comparative study (that included a small subset of patients with eGFR 15-29 mL/min/1.7m2), avacopan was superior to glucocorticoids taper with respect to sustained remission at week 52. In the avacopan arm, the cumulative dose of GCs was dramatically reduced and avacopan was thus proposed as an alternative to GCs rather to a synergic treatment. In the subgroup of patients with eGFR <30 mL/min/1.73m², avacopan was associated with a better eGFR gain at week 52 compared to prednisone, but data in this population at-risk of worse kidney outcomes are scarce, and did not include patients with eGFR < 15 mL/min/1.73m², those patients being excluded from the study.

In the REVERSE study, investigators put forward the hypothesis that avacopan added on GCs regimen may significantly improve the kidney outcome of severe AAV (synergic approach), and thus improve short- and long-term global outcomes (survival, cardiovascular status). REVERSE will thus compare GCs-based SOC + placebo to GCs-based SOC + avacopan.

ELIGIBILITY:
Inclusion Criteria:

* Kidney biopsy before inclusion available (up to 6 weeks before inclusion) or patients agreeing to have a renal biopsy procedure performed no later than prior the visit at week 4
* Have been newly diagnosed or relapsing active AAV-related RPGN at the time of inclusion (either granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA), according to the American College of Rheumatology/European League Against Rheumatism 2022 (ACR/EULAR 2022) classification criteria, with or without positive ANCA testing)
* Have an active disease (BVAS ≥ 3, with at least one of the 2 renal items of proteinuria (urinary proteinuria/creatininuria > 300 mg/g) and haematuria (>10 RBC/hpf) within the BVAS), and eGFR 0-29 mL/min/1.7 m2 at inclusion
* Be planned to receive a SOC induction regimen by rituximab or cyclophosphamide plus glucocorticoids (+ or - plasma exchanges) for the current AAV flare (rituximab or cyclophosphamide may have been started before the inclusion in the study, maximum 2 weeks before the inclusion)
* Affiliated person or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator
* For women able to procreate, ongoing effective contraception

Exclusion Criteria:

* • Irreversible medical conditions likely to affect short-term survival or ability to participate in the study protocol

  * Treatment by >3000 mg methylprednisolone or equivalent within the 3 weeks preceding the screening visit
  * Known eGFR before the AAV flare already <35 mL/min/1.73m2
  * Glomerulosclerosis >60% or kidney interstitial fibrosis >60%, if results of a kidney biopsy are available. If kidney biopsy is performed after inclusion in the study, the patients will continue the study according to the protocol whatever the extent of glomerulosclerosis or interstitial fibrosis.
  * Pregnant or breast-feeding women, or desire to become pregnant within 24 months. All women of childbearing potential (WOCBP) are required to have a negative pregnancy test before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using an effective method of birth control from the date of consent through the end of the study and another 12 months after (or 12 months after the last rituximab infusion in case of premature termination): Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (Oral, Intravaginal, Transdermal); Progestogen-only hormonal contraception associated with inhibition of ovulation (Oral, Injectable, Implantable); Intrauterine device (IUD); Intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomised partner.
  * Hepatic dysfunction defined as:

ALT,AST or alkaline phosphatase > 3 ×ULN Total Bilirubin >2 × ULN, with the exception of participants with Gilbert syndrome who may be included if their total bilirubin is ≤ 3.0 × ULN and direct bilirubin ≤ 1.5 × ULN International normalized ratio (INR) >1.7 (excepted if patient receive vitamin K antagonists)

* Patients with leukocytes below 2000/mm3 or neutrophils below 1000/mm3 will be excluded. However, since patients may have received rituximab or cyclophosphamide before inclusion as a part of induction regimen of the AAV (see inclusion criteria), and both are considered as lymphodepleting agent, mild to moderate lymphopenia (400 - 1500/mm3) at randomization will be allowed
* Co-administration of strong CYP3A4 enzyme inducers
* Known allergy to avacopan
* Other clinically active systemic autoimmune disease requiring therapy, including but not limited to: eosinophilic granulomatosis with polyangiitis (EGPA), moderate to severe systemic lupus erythematosus, IgA vasculitis (Henoch-Schönlein), rheumatoid vasculitis, Sjögren's syndrome, cryoglobulinemic vasculitis, autoimmune hemolytic anemia, autoimmune lymphoproliferative syndrome or mixed connective tissue disease.
* Human immunodeficiency virus (HIV) positivity.
* Acute or chronic infection with hepatitis B (HBV) or hepatitis C (HCV).
* Positive serology for hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg) excludes the participant regardless of detection of hepatitis B surface antibodies (HBsAb) or HBV-DNA.
* Participants with a positive HCV antibody test should have HCV ribonucleic acid (RNA) levels measured. Participants with positive (detectable) HCV RNA must be excluded. Chronic hepatitis C participants, who have completed anti- HCV treatment for at least 12 weeks must have a negative HCV RNA result before randomization. Cases of spontaneous HCV clearance should be discussed with sponsor before enrolment.
* Active viral, bacterial or other infections requiring systemic treatment, or history of recurrent clinically significant infection which in the opinion of the investigator will place the participant at risk for participation.
* Uncontrolled diabetes mellitus, lung diseases or any other illnesses not related to GPA/ MPA that in the opinion of the Investigator would jeopardize the ability of the patient to tolerate glucocorticoids
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 3 years (except for basal cell carcinoma or actinic keratosis that have been treated with no evidence of recurrence in the past 3 months, carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
* Severe heart failure history (i.e., LVEF < 30%)
* Solid organ transplantation
* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations.
* Patient under legal protection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in the kidney function | Day 0 and 52 weeks after randomization
  Proportion of patients reaching an estimated glomerular filtration rate > or = 30 mL/min/1.7m² (CKD-EPI formula applied to the measure of standardized serum creatinine) at week 52 without requiring treatment study discontinuation for serious adverse event or treatment modification or intensification for refractory vasculitis or relapse.

SECONDARY OUTCOMES:
Survival in both groups | Day 0, 52 and 64 weeks after randomization
  percentage of patients alive (and Kaplan Meier survival curves)
Assessment of vasculitis activity | Day 0, 20, 52 and 64 weeks after randomization
  The vasculitis activity is a composite measure derived from Birmingham Vasculitis Activity Score (BVAS; evaluation at weeks 0, 20, 52, 64) and Vasculitis Damage Index (change between baseline (week 0) and weeks 20, 52 and 64, respectively)
Assessment of kidney function | Day 0, 20, 52 and 64 weeks after randomization
  The kidney function is a composite measure derived from changes in eGFR from baseline (in mL/min/1.7m2; CKD-EPI formula derived from the serum creatinine) and Urinary protein/creatinine ratio (mg/mmol) and urinary albumin/creatinine ratio (mg/mmol)
the proportion of end-stage kidney disease | Day 0, 20, 52 and 64 weeks after randomization
  the proportion of end-stage kidney disease is a composite measure derived from number and % percentage ofpatients requiring chronic dialysis
the evolution of the kidney inflammation | Day 0, 4, 12, and 52 weeks after randomization
  the evolution of the kidney inflammation is a composite measure derived from urinary levels of MCP-1 and soluble CD163 and urinary and serum levels of C3a, C5a and factor Bb
Changes in quality of life | Day 0 and 64 weeks after randomization
  Changes in quality of life is a composite measure derived from Short Form-36 component and domain scores and the EuroQOL-5D-5L visual analogue scale (in mm) and index
The assessment the ability of kidney biopsy results to predict the renal response to avacopan | Day 0, 20 and 52 weeks after randomization
  The ability of kidney biopsy results to predict the renal response to avacopan is measured and defined as eGFR ≥ 30mL/min/1.73m2
Safety of treatment | Day 0 and 64 weeks after randomization
  Percentage of patients reporting infections, diabetes mellitus, hepatitis and other adverse events

CONTACTS AND LOCATIONS:
Locations (30):
- France (30):
  - Amiens Hospital, Amiens
  - Angers Hospital, Angers
  - Besançon Hospital, Besançon
  - Bordeaux Hospital, Bordeaux
  - Boulogne-sur-Mer Hospital, Boulogne-sur-Mer
  - Brest Hospital, Brest
  - Caen Hospital, Caen
  - Grenoble Hospital, Grenoble
  - Vendée Hospital, La Roche-sur-Yon
  - Le Mans Hospital, Le Mans
  - Lille Hospital, Lille
  - Limoges Hospital, Limoges
  - Marseille Hospital, Marseille
  - Nantes Hospital, Nantes
  - Nimes Hospital, Nîmes
  - Bichat Hospital, Paris
  - Cochin Hospital, Paris
  - George Pompidou Hospital, Paris
  - Henri Mondor Hospital, Paris
  - Kremlin Bicêtre Hospital, Paris
  - Necker Hospital, Paris
  - Tenon Hospital, Paris
  - Reims Hospital, Reims
  - ROuen Hospital, Rouen
  - Strasbourg Hospital, Strasbourg
  - Saint exupery hospital, Toulouse
  - Toulouse Hospital, Toulouse
  - Tours Hospital, Tours
  - Valenciennes Hospital, Valenciennes
  - NANCY Hospital, Vandœuvre-lès-Nancy